CLINICAL TRIAL: NCT06732011
Title: Evaluation of Brain Dysfunction in Patients with Duchene Muscular Dystrophy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Hassan Ibrahim Ibrahim, Resident doctor, Assiut University
Other Study IDs: Brain evaluation in duchenne
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; Brain; Evaluation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To study the cognitive function & psychiatric aspects of patients with DMD by specific psychometry tests & its relation to quality of life of the patients To evaluate brain structural changes using MRI and correlate them to the cognitive & psychiatric manifestations of the patients To correlate the cognitive function with the neurophysiological tests and imaging done to the patient

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the second most common inherited genetic disease. It is an X-linked disease that affects approximately one in 3300 live male birth. It is caused by the absence or disruption of the dystrophin protein that is a main component of the dystrophin-glycoprotein complex (DGC). It is found in a variety of tissues, mostly skeletal muscle and neuron cells in specific regions of the CNS ashippocampus, the cerebellum and the neocortex. [1, 2] Clinically DMD is characterized by a severe pathology of the skeletal musculature that results in progressive weakness of muscles including cardiac & respiratory muscles leading to the premature death of the individual.

An important aspect of DMD is the neurocognitive function of patients which, despite its non-progressive nature, still greatly affects the quality of life of the patients and their caregivers.[3]

While not all patients exhibit global cognitive impairments, many do show significant deficits in areas such as arithmetic, verbal fluency, working memory, attention, and executive function. A study by Wingeier et al. (2011) found that boys with DMD scored lower than average on IQ tests, particularly in verbal IQ. Other studies have linked specific cognitive impairments to the absence of certain dystrophin isoforms suggesting a genotype-phenotype correlation between mutation and brain affection, particularly Dp140 and Dp260, which are associated with learning disabilities, ADHD, and autism spectrum disorders (ASD).[1, 3, 4]

Many DMD patients face learning difficulties like those seen in developmental dyslexia, this was attributed to the potential role of cerebellar dysfunction & choline deficit in these cognitive dysfunctions, suggesting that metabolic abnormalities in the cerebellum may contribute to the observed impairments. Overall, the research findings emphasize the need for early intervention and highlight the complex interplay of genetic and non-genetic factors in cognitive function among DMD patients.[5-8]

Neuroimaging studies have revealed structural and functional brain abnormalities, with MR spectroscopy and PET showing metabolic abnormalities. Evidence is also emerging for brain regional volume loss, blood oxygen level-dependent signal abnormalities, and altered WM integrity as measured using Diffusion Tensor Imaging. Furthermore, recent imaging studies have highlighted less severe structural abnormalities in patients with retained Dp140 expression compared with those lacking it.[9-11]

ELIGIBILITY:
Inclusion Criteria:

- Male patients Age children & adolescent (5-18yrs) Patients diagnosed & genetically confirmed DMD, with cross matching of healthy subjects of the same age and number

Exclusion Criteria:

Medical or neurological condition affecting cognition (as endocrinal as Diabetes Mellitus & hypothyroidism, autoimmune disease, history of brain trauma, birth asphyxia, neonatal jaundice, …..) Surgical condition that could potentially impact cognitive function Patients of other types of muscular dystrophy Those who refuse to participate in the study Those with sensory disability (as hearing loss, blindness, severe speech delay) Those with non-invasive or invasive ventilation support with inability to speak and answer oral questions

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male
Study Population: Children
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Screening for early detection and management | 2 years